CLINICAL TRIAL: NCT06870513
Title: Comparative Study Between Antegrade and Retrograde Cerebral Perfusion in Acute or Subacute Aortic Dissection Type (A) Patients
Brief Title: Comparative Study of Antegrade Versus Retrograde Cerebral Perfusion in Acute Type A Aortic Dissection: A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yusuf Shieba (Other)
Responsible Party: Sponsor-Investigator, Yusuf Shieba, DR, South Valley University
Organization: South Valley University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCU-FOM-CTS-2020-4222
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Acute Type A Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antegrade cerebral perfusion (ACP) (Experimental): Participants underwent surgical repair of acute Type A aortic dissection utilizing antegrade cerebral perfusion. The procedure involved right axillary artery cannulation through an interposition conduit graft (7-mm Dacron tube) for cardiopulmonary bypass and cerebral perfusion during deep hypothermic circulatory arrest (DHCA).
  Interventions: Procedure: Antegrade Cerebral Perfusion via Axillary Artery
- Retrograde Cerebral Perfusion (RCP) (Active Comparator): Participants in this arm underwent surgical repair of acute Type A aortic dissection utilizing retrograde cerebral perfusion (RCP). Perfusion was provided retrogradely via superior vena cava (SVC) cannulation during deep hypothermic circulatory arrest (DHCA).
  Interventions: Procedure: Retrograde Cerebral Perfusion via Superior Vena Cava

INTERVENTIONS:
Procedure: Antegrade Cerebral Perfusion via Axillary Artery — In antegrade cerebral perfusion (ACP), patients underwent cannulation of the right axillary artery using an interposition Dacron graft (7 mm) connected to a cardiopulmonary bypass (CPB) circuit. During surgery, ACP delivered oxygenated blood flow directly into the brain arteries to maintain cerebral protection during the period of deep hypothermic circulatory arrest (DHCA), enabling the surgical team to perform the distal aortic anastomosis safely.
  Other Names: Antegrade Brain Perfusion
  Arms: Antegrade cerebral perfusion (ACP)
Procedure: Retrograde Cerebral Perfusion via Superior Vena Cava — In retrograde cerebral perfusion (RCP), cannulation of the superior vena cava (SVC) was performed to deliver blood flow in reverse direction during deep hypothermic circulatory arrest (DHCA). This method aimed to provide cerebral protection by supporting cerebral metabolism during the surgical repair of acute Type A aortic dissection.
  Other Names: Retrograde Brain Perfusion
  Arms: Retrograde Cerebral Perfusion (RCP)

SUMMARY:
This prospective study investigated the comparison of effectiveness of antegrade cerebral perfusion (ACP) and retrograde cerebral perfusion (RCP) in providing cerebral protection during the surgical treatment of acute Type A aortic dissection (TAAD). Acute type A aortic dissection presents an aortic tear at its ascending portion, posing considerable risk with high morbidity and mortality incidence, especially from neurological insults.

In total, 116 patients with acute type A aortic dissection were randomly assigned to undergo surgical intervention with either ACP through axillary artery cannulation or RCP through superior vena cava cannula placed during deep hypothermic circulatory arrest. Primary objectives focused on measuring and comparing the postoperative neurological complication rates associated with transient neurological deficits (TND) and permanent neurological deficits (PND). Secondary outcomes of interest included the duration of mechanical ventilation, length of stay in the ICU and hospital, and mortality.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with acute type A aortic dissection (TAAD).

Exclusion Criteria:

* Hemodynamic instability.
* Known ischemic heart disease (IHD).
* History of cerebrovascular stroke.
* Heart failure.
* Renal or hepatic impairment.
* Rheumatic heart disease.
* Previous history of radiotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Neurological Complications (Transient and Permanent Neurological Deficits) | Postoperative assessment period (up to 30 days after surgery)
  Comparison of the incidence of neurological complications, including transient neurological deficits (temporary postoperative mental status changes or neurological dysfunction resolving within 24 hours) and permanent neurological deficits (lasting neurological impairments such as stroke, paralysis, coma, or death).

SECONDARY OUTCOMES:
Postoperative Mortality Rate | 30 days post-surgery
  Comparison of mortality rates within 30 days following surgical intervention between the two perfusion groups (ACP vs. RCP).

CONTACTS AND LOCATIONS:
Overall Officials: Hany Anis Eldomiaty, Professor, Study Chair — Department of Cardiothoracic Surgery, Faculty of Medicine, Suez Canal University, Suez, Egypt.
Locations (1):
- Department of Cardiothoracic Surgery, Faculty of Medicine, Suez Canal University., Suez Canal, Ismailia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to publicly share individual participant data (IPD). Data sharing was not included in the informed consent, and privacy regulations restrict the sharing of individual-level data.

REFERENCES:
- [Background] Samanidis G, Kanakis M, Khoury M, Balanika M, Antoniou T, Giannopoulos N, Stavridis G, Perreas K. Antegrade and Retrograde Cerebral Perfusion During Acute Type A Aortic Dissection Repair in 290 Patients. Heart Lung Circ. 2021 Jul;30(7):1075-1083. doi: 10.1016/j.hlc.2020.12.007. Epub 2021 Jan 22. PMID 33495130
- [Background] Sugiura T, Imoto K, Uchida K, Minami T, Yasuda S. Comparative study of brain protection in ascending aorta replacement for acute type A aortic dissection: retrograde cerebral perfusion versus selective antegrade cerebral perfusion. Gen Thorac Cardiovasc Surg. 2012 Oct;60(10):645-8. doi: 10.1007/s11748-012-0142-z. Epub 2012 Aug 18. PMID 22903579
- [Background] Tokuda Y, Miyata H, Motomura N, Oshima H, Usui A, Takamoto S; Japan Adult Cardiovascular Database Organization. Brain protection during ascending aortic repair for Stanford type A acute aortic dissection surgery. Nationwide analysis in Japan. Circ J. 2014;78(10):2431-8. doi: 10.1253/circj.cj-14-0565. Epub 2014 Aug 28. PMID 25168277
- [Background] Sun S, Chien CY, Fan YF, Wu SJ, Li JY, Tan YH, Hsu KH. Retrograde cerebral perfusion for surgery of type A aortic dissection. Asian J Surg. 2021 Dec;44(12):1529-1534. doi: 10.1016/j.asjsur.2021.03.047. Epub 2021 Apr 20. PMID 33888364
- [Background] Kruger T, Weigang E, Hoffmann I, Blettner M, Aebert H; GERAADA Investigators. Cerebral protection during surgery for acute aortic dissection type A: results of the German Registry for Acute Aortic Dissection Type A (GERAADA). Circulation. 2011 Jul 26;124(4):434-43. doi: 10.1161/CIRCULATIONAHA.110.009282. Epub 2011 Jul 11. PMID 21747050